CLINICAL TRIAL: NCT04371822
Title: Efficacy of Based MRI Contrast Media Against Covid-19
Brief Title: Efficacy of Sunlight Activated Synthetic Porphyrin in COVID-19 Infected Patients
Acronym: SnPPIX
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mahmoud Ramadan mohamed Elkazzaz, Principal Investigator, Kafrelsheikh University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Proposed by Mahmoud Elkazz
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — tin protoporphyrin IX; tetraphenylporphine sulfonate

STUDY DESIGN:
Intervention Model Description: Patients and method :
  This study will performed on 56 participants tested positive for the presence of COVID-19 RNA by RT-PCR kit for RNA detection and 56 participants will divided into 8 equal groups
Masking Description: Patients
  This study will performed on 56 participants tested positive for the presence of COVID-19 RNA by RT-PCR kit for RNA detection and 56 participants will divided into 8 equal groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- 5 mg SnPP dose plus sunlight exposure (Active Comparator): 7 subjects with COVID-19 infection and Serum ferritin < 500 ng/ml will receive a single dose of 5 mg of Stannous Protoporphyrin and They will be exposed to sunlight one hours every day for 14 days
  Interventions: Drug: SnPP Protoporphyrin plus Sunlight exposure
- 7mg SnPP dose plus sunlight exposure (Active Comparator): 7 subjects with COVID-19 infection and Serum ferritin < 500 ng/ml will receive a single dose of 7 mg of Stannous Protoporphyrin and They will be exposed to sunlight two hours every day for 14 days
  Interventions: Drug: SnPP Protoporphyrin plus Sunlight exposure
- 9 mg SnPP dose plus sunlight exposure (Active Comparator): 7 subjects with COVID-19 infection and Serum ferritin < 500 ng/ml will receive a single dose of 9 mg of Stannous Protoporphyrin and They will be exposed to sunlight three hours every day for 14 days
  Interventions: Drug: SnPP Protoporphyrin plus Sunlight exposure
- 5mg TPPS dose plus sunlight exposure (Active Comparator): 7 subjects with COVID-19 infection and Serum ferritin < 500 ng/ml will receive a single dose of 5 mg of sulfonatoporphyrin(TPPS), and They will be exposed to sunlight two hours every day for 14 days
  Interventions: Drug: Sulfonatoporphyrin(TPPS) plus Sunlight exposure.
- placebo (Placebo Comparator): No intervention
  Interventions: Other: placebo

INTERVENTIONS:
Drug: SnPP Protoporphyrin plus Sunlight exposure — SnPP Protoporphyrin plus Sunlight exposure
  Other Names: SnPP
  Arms: 5 mg SnPP dose plus sunlight exposure
Drug: SnPP Protoporphyrin plus Sunlight exposure — SnPP Protoporphyrin and Sunlight exposure
  Other Names: SnPP
  Arms: 7mg SnPP dose plus sunlight exposure
Drug: SnPP Protoporphyrin plus Sunlight exposure — SnPP Protoporphyrin plus Sunlight exposure
  Arms: 9 mg SnPP dose plus sunlight exposure
Drug: Sulfonatoporphyrin(TPPS) plus Sunlight exposure. — Sulfonatoporphyrin(TPPS) plus Sunlight exposure.
  Other Names: (TPPS)
  Arms: 5mg TPPS dose plus sunlight exposure
Other: placebo — No Intervention
  Arms: placebo

SUMMARY:
Efficacy of Sunlight Activated Synthetic Porphyrin in COVID-19 Infected Patients (SnPPIX)

Mahmoud ELkazzaz(1),Rokia yousry abdelaziz sallam(2)

______________________________________________________________________________________________________________________________________________________________________

Abstract :

The novel coronavirus pneumonia (COVID-19) is an infectious acute respiratory caused by the novel coronavirus. The virus is a positive-strand RNA virus with high homology to bat coronavirus. Depending on published study in which , conserved domain analysis, homology modeling, and molecular docking were used to compare the biological roles of specific proteins of the novel coronavirus. The principal investigator demonstrated according to previous researches that some viral structural and nonstructural proteins could bind to the porphyrin, respectively. At the same time, orf1ab, ORF10 and ORF3a proteins coordinated to attack heme on the 1-beta chain of hemoglobin, COVID-19 binds to the porphyrin of haem and displaces iron and a study denonestrated that Covid-19 could cause acquired acute porphyria which is the condition in which there is excess accumulation of porphyrin intermediate metabolites. This point can be taken advantage of X-ray induced visible luminescence of porphyrin for producing of Reactive Oxygen Species (ROS).Many porphyrins are benign in the dark but are transformed by sunlight into caustic, flesh-eating toxins Porphyrins have been used for photodynamic therapy (PDT) against a wide range of targets like bacteria, viruses and tumor cells It has been reported that ROS-based inactivation of viruses may occur due to several reasons, such as protein oxidation, single strand breaks in the RNA genome and protein-RNA crosslinking. Since ROS-based inactivation has a multi-targeted mechanism, it is much less likely that a virus would be able to develop resistance against it. Recently, porphyrins, already in use as photosensitizers for Photodynamic Therapy (PDT), were a study target to applications in medical area, namely as possible contrast agents in MRI. could be observed some examples of porphyrin derivatives already study as MRI contrast media. Low dark toxicity, neoplastic tissue affinity and synthetic accessibility are some of the important properties that contribute for its selection. In MRI studies was found that CM based on paramagnetic metalloporphyrins showed higher affinity for neoplastic tissues, observed by increased relaxation time of the neoplastic tissues, which is reflected on an increase in MRI signal and consequently in a better neoplastic lesions detection. A study demonestrated that The sulfonated tetranaphthyl porphyrin contrast agents in MRI (TNapPS), sulfonated tetra-anthracenyl porphyrin (TAnthPS), and sulfonated 2,6-difluoro-meso-tetraphenylporphine [TPP(2,6-F2)S] and its copper chelate [TPP(2,6-F2)S,Cu], which reduced HIV infection by 99, 96, 94, and 96%, respectively. Previous studies which showed that Covid -19 binds to the porphyrin of haem and displaces iron in addition to Sulfonated porphyrins and light-stimulated Sn- protoporphyrin IX have broad antiviral activity against more distinct types of viruses, Co-protoporphyrin IX and Sn-protoporphyrin IX inactivate Zika, Chikungunya and other arboviruses by targeting the viral envelope Porphyrins are amphipathic molecules able to interact with membranes and absorb light, being widely used in photodynamic therapy. Previously, we showed that heme, Co-protoporphyrin IX (CoPPIX) and Sn-protoporphyrin IX (SnPPIX) directly inactivate DENV and YFV infectious particles. Here we demonstrate that the antiviral activity of these porphyrins can be broadened to CHIKV, ZIKV, Mayaro virus, Sindb is virus and Vesicular Stomatitis virus. Porphyrin treatment causes viral envelope protein loss, affecting viral morphology, adsorption and entry into target cells , Finally, the principal investigator expect that viral load will be declined with sunlight because In particular, porphyrins absorb essentially all the UV/visible light wavelengths in the emission spectrum of the sun; hence they are active at very low doses .

Keywords: COVID 2019 ,Infection, Sulfonated porphyrins and X-ray induced visible luminescence of porphyrin

DETAILED DESCRIPTION:
Efficacy of Sunlight Activated Synthetic Porphyrin in COVID-19 Infected Patients (SnPPIX)

Official Title: Efficacy of Based MRI Contrast Media Against Covid-19

____________________________________________________________________________________________________________________________________________________________

Introduction:

Pandemic Covid-19 pneumonia, of SARS-CoV-2 aetiology, presents an existential threat to health care systems globally. Multiple therapeutic and prophylactic agents are currently undergoing clinical trial, including 23 clinical trials of (hydroxy) chloroquine in China. While progress towards a curative agent or vaccine is promising, the principal limiting factor in public health emergency is time, and therefore Virus resistance to antiviral therapies is an increasing concern that makes the development of broad-spectrum antiviral drugs urgent. Targeting of the viral envelope, a component shared by a large number of viruses, emerges as a promising strategy to overcome this problem. Natural and synthetic porphyrins are good candidates for antiviral development due to their relative hydrophobicity and pro-oxidant character a pre-existing licensed therapeutic would offer reprieve to health care systems operating at the edge of capacity. In this brief communication, the Principal investigator argues that Covid-19 has high probability of being more than a disease of pneumonia, and that critical Covid-19 patients may be experiencing a form of acquired acute porphyria. Readily available interventions exist to treat acute porphyria and the position is advanced that urinalysis of critical Covid-19 patients would diagnose this pathology.

COVID-19 binds to porphyrin and cause acquired porphyria.

Erythrocytes are strongly implicated in the pathophysiology of Covid-19. Wuhan University researchers argue that the role of erythrocytes in the pathophysiology of Covid-19 is under-estimated; the co-efficient of variation of red blood cell distribution width (RDW) is predictive of severity of disease state (Gong 2020). Elevated RDW is correlated with reduced erythrocyte turnover; red blood cells become smaller as they age and the delay in clearance expands the low-volume tail of the volume distribution (Patel 2015). Suppressed erythrocyte turnover may indicate erythropoietic distress and function as a compensatory mechanism to maintain circulating red blood cell levels (Patel 2015).

Excess porphyrins in red blood cells can precipitate cell lysis and development of hemolytic anaemia (Sassa 2006). Macaques infected with SARS-CoV- 2 also have decreased red blood cell numbers (Munster 2020) and susceptibility to SARS-CoV-2 appears to be determined by blood group; blood group A is most affected whereas blood group O seems to be protected (Yang 2020). This finding is concordant with previous studies showing that susceptibility to the 2003 strain of SARS-CoV was determined by blood group (Guillon 2008). Preliminary evidence suggests that CD147, the determinant of the Ok blood group system, binds the spike protein of SARS-CoV-2 (Wang 2020). Incidentally, CD147 functions as an essential receptor for erythrocyte invasion by Plasmodium falciparum (Crosnier 2011). Blockade of CD147 abrogates the normal recirculation of erythrocytes, from the spleen into the general circulation, leading to selective trapping of red blood cells in the spleen as development of a form of anaemia (Coste 2001). Autopsy of deceased Covid-19 patients reveals that the spleen is significantly reduced in size. Reduction in spleen size would be expected in the event that the spleen has emptied its reserve of erythrocytes into the circulation as part of a normal physiological response to anaemia (Dale 2016).

Primate models of Covid-19 (Munster 2020) and human Covid-19 patients have subnormal haemoglobin levels (Chen 2020). Clinical evaluation of almost 100 Wuhan patients reveals haemoglobin levels below the normal range in most patients as well as increased total bilirubin and elevated serum ferritin (Chen 2020). Hyperbilirubinemia is observed in acute porphyria (Sassa 2006) and would be consistent with ineffective erythropoiesis (Sulovska 2016) and rapid haemoglobin turnover.

COVID-19 and Porphyrin of haem:-

Elevated serum ferritin levels are typical of acute porphyria (Trier 2013) and would be expected upon dissociation of iron from haem. A mechanism by which SARS-CoV-2 might attack the 1beta chain of haemoglobin has been proposed; the product of open reading frame 8 (ORF8) binds to the porphyrin of haem and displaces iron, according to bioinformatics prediction analyses (Liu 2020).

The oxygen-carrying capacity of erythrocytes would therefore be compromised by SARS-CoV-2, thereby exacerbating the difficulties already experienced by the patient, in terms of maintaining partial pressure of oxygen in the alveoli (PaO2). While the impact of SARS-CoV-2 targeting of haemoglobin on oxygen content of the blood would therefore be considerable, the author proposes that perhaps of greater concern, are potential ramifications upon homeostatic regulation of haem anabolism. Haem biosynthesis is exquisitely controlled by seven enzyme-controlled reactions proceeding from the first intermediate, aminolevulinic acid (ALA), to haem as thefinal product. Haem negatively regulates the first step in the pathway by repressing expression of aminolevulinic acid synthase (ALAS).

SARSCoV- 2 is predicted to directly interfere with haem production (Liu 2020), and this prediction is supported by empirical evidence of reduced haemoglobin levels in Covid-19 patients (Chen 2020) and in animal models of the disease (Munster 2020). Decreased haem production dampens repression of ALAS, and thereby increases the production of haem precursors, leading to accumulation of porphyrin intermediate metabolites. All of the haem pathway intermediates are potentially toxic (Sassa 2006). During an attack of acute porphyria, ALAS is induced 2006) and this perturbation continues until sufficient haem synthesis is restored. Phenotype of SARS-CoV-2 porphyrin excess is hypothesised to mimic extreme lead poisoning; both as examples of acquired acute porphyria.

Overproduction of haem precursors - aminolevulinic acid (ALA) and porphobilinogen (PBG), in particular - manifests life-threatening attacks (Pischik 2015) with neurovisceral symptoms (Sassa 2006), including: abdominal pain (85-95% cases), vomiting (43-88%), constipation (48-84%), muscle weakness (42-60%), mental symptoms (40-58%), pain of the limbs, head, neck and chest (50-52%), hypertension (36-54%), tachycardia (28-80%), convulsion (10-20%), sensory loss (9-38%), fever (9-37%), respiratory paralysis (5-12%) and diarrhoea (5-12%). Neurotoxicity of aminolevulinic acid accounts for the plethora of neurovisceral symptoms and, interestingly, there is considerable overlap between neurovisceral complaints of ALA excess and extra-pulmonary symptoms of critical Covid-19 patients. Extra-pulmonary symptoms of Covid-19 are significant but under-estimated, including gastrointestinal symptoms (Poggiali 2020), which news reports suggest may affect in the region of 50% Covid-19 patients. Neurological problems also appear to be overlooked by the hyper-focus on respiratory symptoms (Zhao 2020). Of 214 Covid-19 patients, 36.4% experienced neurological manifestations including: headache, dizziness, acute cerebrovascular incidents and impaired consciousness (Mao 2020). Loss of autonomic control of breathing has also been reported and autonomic neuropathy is a clinical feature of acute porphyria (Laiwah 1985). Neuropsychiatric symptoms of Covid-19 may be downstream of irregularities in haem metabolism.

The most important question is now asked by Principal investigator Can Sunlight stimulated porphyrins act against COVID-19 as like as Sn- protoporphyrin IX mechanism in impeding the entry and division of the virus(Zika, Chikungunya and other arbo viruses) by targeting the viral envelope and protect hemoglobin and blood components that are affected by the viral infection?

The principal investigator expect the possibility of inhibiting Covid -19 by Sulfonated porphyrins X-ray induced visible luminescence of porphyrin and light-stimulated Sn- protoporphyrin IX because According to previous studies which showed that Covid -19 binds to the porphyrin of haem and displaces iron in addition to Sulfonated porphyrins and light-stimulated Sn- protoporphyrin IX have broad antiviral activity against more distinct types of viruses, Co-protoporphyrin IX and Sn-protoporphyrin IX inactivate Zika, Chikungunya and other arboviruses by targeting the viral envelope Porphyrins are amphipathic molecules able to interact with membranes and absorb light, being widely used in photodynamic therapy. Previously, we showed that heme, Co-protoporphyrin IX (CoPPIX) and Sn-protoporphyrin IX (SnPPIX) directly inactivate DENV and YFV infectious particles. Here we demonstrate that the antiviral activity of these porphyrins can be broadened to CHIKV, ZIKV, Mayaro virus, Sindb is virus and Vesicular Stomatitis virus. Porphyrin treatment causes viral envelope protein loss, affecting viral morphology, adsorption and entry into target cells (Neris 2018)

The sulfonated tetranaphthyl porphyrin (TNapPS), sulfonated tetra-anthracenyl porphyrin (TAnthPS), and sulfonated 2,6-difluoro-meso-tetraphenylporphine [TPP(2,6-F2)S] and its copper chelate [TPP(2,6-F2)S,Cu], which reduced HIV infection by 99, 96, 94, and 96%, respectively (Andrei 2002)

Treatment of HepG2 cells with heme, CoPPIX and SnPPIX after DENV infection reduced infectious particles without affecting viral RNA contents in infected cells. The reduction of viral load occurs only with the direct contact of DENV with porphyrins, suggesting a direct effect on viral particles. Previously incubation of DENV and YFV with heme, CoPPIX and SnPPIX resulted in viral particles inactivation in a dose-dependent manner. Biliverdin, a noncyclical porphyrin, was unable to inactivate the viruses tested. Infection of HepG2 cells with porphyrin-pretreated DENV2 results in a reduced or abolished viral protein synthesis, RNA replication and cell death. Treatment of HepG2 or THP-1 cell lineage with heme or CoPPIX after DENV infection with a very low MOI resulted in a decreased DENV replication and protection from death. (Assunção 2016)

In summary, SARS-CoV-2 would not be the first known virus to alter porphyrin metabolism; hepatitis C virus (Hep C) and human immunodeficiency virus(HIV) infection lead to a non-acute form of porphyria (Blauvelt 1996). So the principal investigator expects and suggests that porphyrin based therapy is suitable and effective treatment against COVID-19 and could Protects hemoglobin and RBCs from dangerous influence of COVID-19 .The possibility of therapeutic application of porphyrins or their use as models to design new antiviral drugs against DENV ,COVID -19 and YFV.

ELIGIBILITY:
Inclusion Criteria:

Adult SARI patients with 2019-ncov infection confirmed by PCR; Absolute value of lymphocytes < 0. 6x 109/L; Severe respiratory failure within 48 hours and requires admission to ICU. (severe respiratory failure was defined as PaO2/FiO2 < 200 mmHg and was supported by positive pressure mechanical ventilation (including non-invasive and invasive mechanical ventilation, PEEP>=5cmH2O))

Exclusion Criteria:

* History of malignancy except carcinoma in situ in the cervix, early stage prostate cancer or non-melanoma skin cancers. Cancer free for less than 5 years.
* Use of investigational drugs or participation in another clinical trial within 30 days or 5 half-lives prior to screening, whichever is longer.
* Serum ferritin > 500 ng/ml or who have received IV iron within 28 days of screening, or currently being treated with oral iron.
* Women who are pregnant, breastfeeding, or planning to become pregnant while participating in the study.
* Regular use of drugs of abuse and/or positive findings on urinary drug screening.
* Subjects who are severely physically or mentally incapacitated and who, in the opinion of investigator, are unable to perform the subjects' tasks associated with the protocol.
* Presence of any condition which, in the opinion of the investigator, places the subject at undue risk or potentially jeopardizes the quality of the data to be generated.
* Subjects with history of photosensitivity or active skin disease, which, in the opinion of the investigator could increase the risk of photosensitivity.
* Subjects with abnormal baseline liver tests or hepatitis serologies that suggest active infection.
* Liver disease
* Renal disease
* Known hypersensitivity or previous anaphylaxis to SnPP and Sulfonated porphyrins

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
lung injury score | at 7and 14 days
  Proportion of lung injury score decreased or increased after treatment
Serum ferritin | at day 1-3-7 and 14
  Serum ferritin

SECONDARY OUTCOMES:
Absolute lymphocyte counts | at day 7 and 14
  lymphocyte counts
Serum levels of CRP, ESR ,IL-1,IL-6,TNF and Type I interferon | at day 7 and 14
  Serum levels of CRP, ESR ,IL-1,IL-6,TNF and Type I interferon
Serum level of COVID19 RNA | at day 7 and 14
  Serum level of COVID19 RNA
All cause mortality rate | at day 7 and 14
  died
Ventilation free days | at 14 days
  ventilation free days
ICU free days | at 14 days
  ICU free days
d-dimers | at 3-5days
  less than 250 ng/mL, or less than 0.4 mcg/mL of blood sample
Time to first negative SARS-CoV-2 PCR in NP swap | within 14 days
  (if pos. at baseline)

CONTACTS AND LOCATIONS:
Overall Officials: M.Sc. Mahmoud Elkazzaz, M.Sc.in Biochemistry, Study Chair — Damitta University
Locations (1):
- Kafr El-sheikh University, Cairo, Kafr el-Sheikh Governorate, Egypt